CLINICAL TRIAL: NCT01507909
Title: Quantitative EEG Assessment of Cue-Induced Changes in Brain Activity in Alcohol Use Disorders
Status: Terminated | Type: Observational
Why Stopped: Equipment Failure
Sponsor: Boston University (Other)
Responsible Party: Principal Investigator, Ofra Sarid-Segal MD, Medical Director of the Clinical Studies Unit, Boston University
Other Study IDs: EEG CUE study-H-31322
Record Dates: First submitted 2012-01-09; First posted 2012-01-11 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Alcohol Craving
Keywords: EEG; related visual; and verbal cues

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Exposure to alcohol related cues, such as the sight of alcoholic drinks, may induce craving for alcohol in drinkers. In this study, the effects of exposure to (1) the pictures of alcoholic drinks and (2) the imagining of a scene related to drinking on activity in the frontal region of the brain in heavy social drinkers will be determined. This study is being conducted to develop the methods needed to allow for the detection of cue-induced changes in drinkers using the EEG. The objective of this pilot study is to establish procedures for detecting alcohol-related cue-elicited changes in EEG activity in heavy drinkers.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 21 to 70.
2. History of heavy drinking: Defined as at least 8 occasions in the past month that individual had at least 5 drinks (males) or 4 drinks (females) in one sitting.
3. The subject must currently not be in treatment for any alcohol use disorder
4. Subject must be able to comprehend and perform study related information and tasks in English and have a willingness to complete study procedures.
5. Subject must be able to provide written informed consent, at time of consent BAC has to be 0.00%.
6. The subject must have the ability to read/speak English

Exclusion Criteria:

1. Severe impairment of sight, smell, or hearing that would result in a significant alteration in the response to alcohol related cues.
2. Currently on a medication used to treat alcoholism or is known to alter EEG activity or responsiveness to cue presentation including acamprosate, anticonvulsants, anticholinergics, antipsychotics, benzodiazepine receptor agonists, beta adrenergic receptor antagonists, and naltrexone.
3. History of any neurological or psychiatric disorder that would result in abnormal EEG activity such as severe brain trauma, seizure disorders, stroke or that would severly alter response to the cue presentation such as schizophrenia or any other psychotic or severe mood disorder.
4. CIWA-AR score of 8 or higher or any history indicating that the subject is at risk for experiencing severe alcohol withdrawal symptoms if her or his drinking is discontinued for any period of time.
5. The subject must not be pregnant. -

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Local participants not interested in alcohol treatment.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2012-01; Primary Completion 2014-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
FFT power of five frequency bands
  This study will look at FFT power of five frequency bands. Relative power will be determined by finding absolute power for the range of frequencies (0,1 to 100Hz). Relative power will then be found for each electrode. The Investigator's will examine change over time for relative power for each electrode in the different cue condition and compare change of power using repeated measures analysis with time and condition as within subject factors. Craving values obtained under the different cue conditions will be analyzed using condition as the within-subject factor.

CONTACTS AND LOCATIONS:
Overall Officials: Ofra Sarid-Segal, MD, Principal Investigator — Boston University
Locations (1):
- Boston University Medical Center, Boston, Massachusetts, United States